CLINICAL TRIAL: NCT00492986
Title: An Open Label, Non Comparative, Phase III Study of the Raf Kinase Inhibitor BAY 43-9006 as a Subsequent to First Line Therapy in Patients With Advanced Renal Cell Carcinoma
Brief Title: An Open-Label, Non-Comparative, Phase III Study of the Raf-Kinase Inhibitor BAY 43-9006 as a Subsequent to First-Line Therapy in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11941; 2005-002524-34 (EudraCT Number)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Cancer (RCC); Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Multikinase inhibitor: Sorafenib mono therapy 400 mg bid

SUMMARY:
Purpose of the study:

The purpose of this study is to make sorafenib available for patients with advanced Renal Cell Carcinoma, who have failed prior systemic therapy for advanced disease (i.e. requiring second line treatment), and who do not have access to or are not eligible for other clinical trials with sorafenib and who may benefit from treatment with sorafenib.

Patients will be treated orally with 400 mg bid sorafenib on a continuous basis and as a single agent. Patients may continue treatment until Disease Progression, intolerable toxicity, the patients chooses to withdraw consent or the patient is unlikely to benefit any further from treatment.

Overall, participation in the study will help determine the following:

* Find out if patients receiving Sorafenib will live longer
* Find out if Sorafenib helps to slow the worsening of kidney cancer
* Find out if Sorafenib has an effect on the tumours

ELIGIBILITY:
Inclusion Criteria:

* The patient must provide written informed consent prior to receiving BAY 43-9006
* The male or female patient must be at least 18 years of age
* The patient must have advanced Renal Cell Carcinoma
* The patient must have failed at least one prior systemic established therapy for advanced RCC (e. g. IL-2, IFN-a), or must have been unable to tolerate systemic therapy for advanced RCC, or is deemed by the Investigator to be unsuited for systemic therapy for advanced RCC
* A patient, who has received prior systemic and local therapies, must have completely recovered from acute toxicity (i. e. resolved back to CTCAE Grade 1 or less, or is considered as not going to resolve), if any, prior to study entry
* The patient must be, in the Investigator's opinion, reasonably likely to benefit from treatment with BAY 43-9006 as a single agent
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* The patient will not require other systemic anti-cancer chemotherapy, immunotherapy (including monoclonal antibodies) or hormonal therapy, except for bisphosphonates while taking BAY 43-9006
* Both male and female patients must use adequate barrier birth control methods (oral contraceptives, injectable contraceptives, intrauterine devices, condoms, sterilization) during their participation in the protocol. The birth control methods must be used for 4 weeks for female patients and for 3 months for male patients after discontinuation of treatment with sorafenib
* For patients, who have had major surgery, the wound must be completely healed prior to receiving BAY 43-9006 treatment (4 weeks)

Exclusion Criteria:

* Patients who are currently enrolled in or have previously participated in any other sorafenib trial
* Patients, who are eligible for or do have access to any other sorafenib clinical trial as to the knowledge of the Investigator
* Patients who have a life expectancy of less than 2 months
* Patients with metastatic brain or meningeal tumors
* Patients are excluded who require any of the following:
* Investigational drug therapy during the treatment with sorafenib or within 30 days prior to their first dose of sorafenib
* Concomitant Rifampicin
* Concomitant St. John's Wort (Hypericum perforatum) Warfarin is allowed; however, for patients receiving concomitant warfarin therapy close monitoring of Prothrombin Time (PT) should be performed (please note that no laboratory data are collected in this study)
* Women who are pregnant or breast-feeding. Women of childbearing potential must have a negative pregnancy test performed within seven days of the start of study drug (please note that no laboratory data are collected in this study)
* Patients with congestive heart failure greater than NYHA functional class II (symptomatic during ordinary activity)
* Patients with cardiac arrhythmias greater than Grade 1 NCI CTCAE, Version 3.0 (conduction abnormality and supraventricular arrhythmia present but patient is asymptomatic; intervention not indicated, palpitations present and QTc > 0.45-0.47 second)
* Patients with active coronary artery disease or ischemia
* Patients with Child-Pugh class C hepatic impairment
* Patients with severe renal impairment (calculated creatinine clearance of < 30 ml/min) or who require dialysis
* Patients with active uncontrolled hypertension
* Patients with recent or active bleeding diathesis
* Patients with any medical condition which could jeopardize their safety while taking an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Safety Parameters | Continously

SECONDARY OUTCOMES:
Collection of radiological evaluations | Continously

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Århus C, Denmark
- France (3):
  - Bordeaux
  - Lyon
  - Villejuif
- Germany (10):
  - München, Bavaria
  - Hamburg, Hamburg
  - Darmstadt, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Koblenz, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Homburg, Saarland
  - Dresden, Saxony
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
- Italy (5):
  - Milan
  - Modena
  - Pavia
  - Perugia
  - Reggio Emilia
- Amsterdam, Netherlands
- Warsaw, Poland
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
- Sweden (2):
  - Gothenburg
  - Stockholm
- Switzerland (2):
  - Basel, Canton of Basel-City
  - Geneva, Canton of Geneva
- United Kingdom (3):
  - London, London
  - Glasgow, Stratchclyde
  - Sutton, Surrey

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/